CLINICAL TRIAL: NCT04795804
Title: The Effects of Human-like Milk Oligosaccharide and Resistant Starch on Acetate Production and Human Substrate Metabolism
Brief Title: Human Milk Oligossaccharide and Acetate Production in Vivo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NL71611.068.19
Record Dates: First submitted 2020-12-04; First posted 2021-03-12 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-03

CONDITIONS: Obesity; Insulin Resistance
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — maltodextrin; Resistant Starch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): 11.43 g (3 x 3.81 g) maltodextrin the day before the clinical investigation day
  Interventions: Dietary Supplement: Maltodextrin
- Human milk-like oligosaccharide alone (Active Comparator): 12 g (3 x 4 g) of the human milk-like oligosaccharide the day before the clinical investigation day
  Interventions: Dietary Supplement: Human Milk Oligossaccharide
- Human milk-like oligosaccharide and resistant starch (Experimental): 12 g (3 x 4 g) of the human milk-like oligosaccharide and 7.5g resistant starch (3 x 2.5 g) the day before the clinical investigation day
  Interventions: Dietary Supplement: Human Milk Oligossaccharide and resistant starch

INTERVENTIONS:
Dietary Supplement: Human Milk Oligossaccharide — The day before the CIDs, the participants receive the supplements 3x a day in randomized order
  Arms: Human milk-like oligosaccharide alone
Dietary Supplement: Maltodextrin — The day before the CIDs, the participants receive the supplements 3x a day in randomized order
  Arms: Placebo
Dietary Supplement: Human Milk Oligossaccharide and resistant starch — The day before the CIDs, the participants receive the supplements 3x a day in randomized order
  Arms: Human milk-like oligosaccharide and resistant starch

SUMMARY:
The study investigators hypothesize (1) that the SCFA/acetate metabolism differs between metabolic phenotypes and (2) that using a mixture of fibres that differ in degree of polymerization and branching namely a resistant starch and a human-like milk oligosaccharide enhance the acetate availability in the distal colon and systemic circulation, consequently leading to its metabolic effects.

To study this, the investigators will supplement lean, normoglycaemic vs. overweight/obese, prediabetic men with the fibre mixture the day before the clinical investigation day (CID) and study during the CID its effects on fasting and postprandial substrate and energy metabolism.

ELIGIBILITY:
Inclusion criteria:

Lean (BMI ≥ 20kg/m2 and ≤ 24.9kg/m2) healthy men aged 30 - 65 years

as well as

overweight/obese (BMI ≥ 25kg/m2 and ≤ 34.9kg/m2) prediabetic men aged between 30 - 65 years

Exclusion criteria:

* Type 2 diabetes mellitus (defined as fasting plasma glucose ≥ 7.1 mmol/L and 2h glucose ≥ 11.1 mmol/L)
* Gastroenterological diseases or abdominal surgery;
* Cardiovascular diseases, cancer, liver or kidney malfunction, disease with a life expectancy shorter than 5 years;
* Abuse of products; alcohol and drugs, excessive nicotine use defined as >20 cigarettes per day;
* Plans to lose weight or following of a hypocaloric diet;
* Regular supplementation of pre- or probiotic products, use of pre- or probiotics 3 months prior to the start of the study;
* Intensive exercise training more than three hours a week;
* Use of any medication that influences glucose or fat metabolism and inflammation (i.e. NSAIDs);
* Regular use of laxation products;
* Use of antibiotics in the last three months (antibiotics use can alter substantially the gut microbiota composition).
* Follow a vegan diet.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Plasma acetate concentrations. | plasma acetate will be sampled during the CID before the consumption of a liquid high fat mixed meal
  During the clinical investigation day plasma acetate will be sampled
Plasma acetate concentrations. | plasma acetate will be sampled during the CID at t=60 minutes after consumption of a liquid high fat mixed meal
  During the clinical investigation day plasma acetate will be sampled
Plasma acetate concentrations. | plasma acetate will be sampled during the CID at t=120 minutes after consumption of a liquid high fat mixed meal
  During the clinical investigation day plasma acetate will be sampled
Plasma acetate concentrations. | plasma acetate will be sampled during the CID at t=240 minutes after consumption of a liquid high fat mixed meal
  During the clinical investigation day plasma acetate will be sampled
Faecal acetate concentrations. | Fecal acetate will be sampled in the morning before the testday
  On the day of clinical investigation day, fecal acetate will be sampled
Plasma butyrate concentrations. | plasma butyrate will be sampled during the CID before the consumption of a liquid high fat mixed meal
  During the clinical investigation day, plasma butyrate will be sampled
Plasma butyrate concentrations. | plasma butyrate will be sampled during the CID at t=60 after consumption of a liquid high fat mixed meal
  During the clinical investigation day, plasma butyrate will be sampled
Plasma butyrate concentrations. | plasma butyrate will be sampled during the CID at t=120 after consumption of a liquid high fat mixed meal
  During the clinical investigation day, plasma butyrate will be sampled
Plasma butyrate concentrations. | plasma butyrate will be sampled during the CID at t=240 minutes after consumption of a liquid high fat mixed meal
  During the clinical investigation day, plasma butyrate will be sampled
Fecal butyrate concentrations. | Fecal butyrate will be sampled in the morning before the testday
  On the day of clinical investigation day, fecal butyrate will be sampled
Plasma propionate concentrations. | Plasma propionate will be sampled during the CID before the consumption of a liquid high fat mixed meal
  During the clinical investigation day, plasma propionate will be sampled
Plasma propionate concentrations. | Plasma propionate will be sampled during the CID t=60 minutes after the consumption of a liquid high fat mixed meal
  During the clinical investigation day, plasma propionate will be sampled
Plasma propionate concentrations. | Plasma propionate will be sampled during the CID t=120 minutes after the consumption of a liquid high fat mixed meal
  During the clinical investigation day, plasma propionate will be sampled
Plasma propionate concentrations. | Plasma propionate will be sampled during the CID t=240 minutes after the consumption of a liquid high fat mixed meal
  During the clinical investigation day, plasma propionate will be sampled
Faecal propionate concentrations. | Fecal propionate will be sampled in the morning before the testday
  On the day of clinical investigation day, fecal propionate will be sampled

SECONDARY OUTCOMES:
Energy expenditure, fat and carbohydrate oxidation | Indirect calorimetry will be measured before and for 4 hours after the consumption of the liquid high-fat mixed meal during the whole CID
  Energy expenditure, fat and carbohydrate oxidation will be measured using an open-circuit ventilated hood system (Omnical, Maastricht University, The Netherlands);
Breath H2 using (Bedfont EC60 Gastrolyzer, Rochester, UK). | Breath H2 will be sampled during the CID before and at t=30, t=60, t=90, t=120 and t=240 minutes after consumption of a liquid high fat mixed meal
  Breath H2 using (Bedfont EC60 Gastrolyzer, Rochester, UK).
Plasma glucose concentrations | Plasma glucose concentrations will be sampled during the CID before and t=0, t=30, t=60, t=120 and t=240 minutes after consumption of a liquid high fat mixed meal
  Plasma glucose concentrations
Plasma insulin concentrations | Plasma insulin concentrations will be sampled during the CID before and at t=0, t=30, t=60, t=120 and t=240 minutes after consumption of a liquid high fat mixed meal
  Plasma insulin concentrations
Plasma FFA concentrations | Plasma FFA concentrations will be sampled during the CID before and at t=0, t=30, t=60, t=120 and t=240 minutes after consumption of a liquid high fat mixed meal
  Plasma FFA concentrations
Faecal microbiota composition | Faecal microbiota composition will be sampled in the morning before the testday
  Faecal microbiota composition will be assessed via16S rRNA gene sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Canfora EE, Vliex LMM, Wang T, Nauta A, Bouwman FG, Holst JJ, Venema K, Zoetendal EG, Blaak EE. 2'-fucosyllactose alone or combined with resistant starch increases circulating short-chain fatty acids in lean men and men with prediabetes and obesity. Front Nutr. 2023 Jul 17;10:1200645. doi: 10.3389/fnut.2023.1200645. eCollection 2023. PMID 37529001